CLINICAL TRIAL: NCT03201185
Title: Beneficio Del Bloqueo Del Sistema Renina-angiotensina Sobre la evolución clínica y el Remodelado Ventricular Tras la colocación de Una prótesis percutánea aórtica (RASTAVI)
Brief Title: Renin-angiotensin System Blockade Benefits in Clinical Evolution and Ventricular Remodeling After Transcatheter Aortic Valve Implantation (RASTAVI)
Acronym: RASTAVI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Carlos Baladron, PhD, Research Coordinator, Cardiology, Hospital Clínico Universitario de Valladolid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCUValladolid
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Transcatheter Aortic Valve Replacemen; Angiotensin-Converting Enzyme Inhibitors
Keywords: Cardiovascular events; Ventricular remodeling
MeSH Terms: conditions — Ventricular Remodeling | interventions — Ramipril

STUDY DESIGN:
Intervention Model Description: Open-label
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ramipril (Experimental): After transcatheter aortic valve implantation, patients will receive ramipril before discharge plus conventional treatment (in patients without ACEI).
  Interventions: Drug: Ramipril
- No intervention (No Intervention): Conventional treatment after transcatheter aortic valve implantation

INTERVENTIONS:
Drug: Ramipril — Initial dose: 2,5 mg. Up-titrated at one month to 5 mg and 10 mg at three months (following clinical practice recommendations for up-titration). Target dose: 10 mg (or maximum tolerated dose).
  Arms: Ramipril

SUMMARY:
The investigators aim to demonstrate that ramipril after transcatheter aortic valve implantation has benefits in terms of prognosis, cardiovascular events and ventricular remodeling (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Transcatheter aortic valve implantation due to severe aortic stenosis.
* Patients must give written informed consent.

Exclusion Criteria:

* Severe mitral valvulopathy.
* Reduced left ventricular ejection fraction (LVEF < 40%) with myocardial infarction or dilated cardiomyopathy.
* Patients on an ACEI or an ARB the last 3 months.
* History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACEIs, ARBs, or NEP inhibitors as well as known or suspected contraindications to the study drugs.
* Non-MR-conditional cardiac devices.
* Estimated GFR < 30 ml/min. GFR between 30 and 50 ml/min will not receive gadolinium during MRI.
* Systolic blood pressure < 100 mmHg or diastolic < 40 mmHg.
* Pregnant women.
* Participating in other investigational trial at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants that had the occurrence of cardiovascular events (cardiac death, heart failure admission and stroke). | Up to 36 months
  Number of participants that had first occurrence of cardiovascular events, which is defined as either cardiac death or heart failure hospitalization or stroke

SECONDARY OUTCOMES:
Changes in left ventricular remodeling at 12 months assessed by cardiac MRI. Changes in left ventricle ejection fraction, ventricular dimenssions, ventricular mass and myocardial fibrosis will be measured | Up to 12 months
  Myocardial fibrosis will be measured in grams
Change from baseline to month 12 for the six minutes walk test in order to assess functional capacity. | Up to 12 months
  Assessed by six minutes walk test at 12 months
Number of patients dead due to cardiac causes. | Up to 12 and 36 months
  Number of patients dead due to cardiac causes at 12 and 36 months.
Number of patients admitted due to heart failure. | Up to 12 and 36 months
  Number of patients admitted due to heart failure at 12 and 36 months.
Number of patients with stroke (Defined as compatible symptoms or confirmed by imaging technique: MRI or CT) during the trial. | Up to 12 and 36 months
  Number of patients with stroke during the trial at 12 and 36 months.
Number of patients - All-cause mortality | Up to 12 and 36 months
  All-cause mortality measures how many patients had this event at 12 and 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

REFERENCES:
- [Background] Lindroos M, Kupari M, Heikkila J, Tilvis R. Prevalence of aortic valve abnormalities in the elderly: an echocardiographic study of a random population sample. J Am Coll Cardiol. 1993 Apr;21(5):1220-5. doi: 10.1016/0735-1097(93)90249-z. PMID 8459080
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Background] Del Trigo M, Munoz-Garcia AJ, Wijeysundera HC, Nombela-Franco L, Cheema AN, Gutierrez E, Serra V, Kefer J, Amat-Santos IJ, Benitez LM, Mewa J, Jimenez-Quevedo P, Alnasser S, Garcia Del Blanco B, Dager A, Abdul-Jawad Altisent O, Puri R, Campelo-Parada F, Dahou A, Paradis JM, Dumont E, Pibarot P, Rodes-Cabau J. Incidence, Timing, and Predictors of Valve Hemodynamic Deterioration After Transcatheter Aortic Valve Replacement: Multicenter Registry. J Am Coll Cardiol. 2016 Feb 16;67(6):644-655. doi: 10.1016/j.jacc.2015.10.097. PMID 26868689
- [Background] Cioffi G, Faggiano P, Vizzardi E, Tarantini L, Cramariuc D, Gerdts E, de Simone G. Prognostic effect of inappropriately high left ventricular mass in asymptomatic severe aortic stenosis. Heart. 2011 Feb;97(4):301-7. doi: 10.1136/hrt.2010.192997. Epub 2010 Aug 18. PMID 20720251
- [Background] Dweck MR, Joshi S, Murigu T, Alpendurada F, Jabbour A, Melina G, Banya W, Gulati A, Roussin I, Raza S, Prasad NA, Wage R, Quarto C, Angeloni E, Refice S, Sheppard M, Cook SA, Kilner PJ, Pennell DJ, Newby DE, Mohiaddin RH, Pepper J, Prasad SK. Midwall fibrosis is an independent predictor of mortality in patients with aortic stenosis. J Am Coll Cardiol. 2011 Sep 13;58(12):1271-9. doi: 10.1016/j.jacc.2011.03.064. PMID 21903062
- [Background] Schunkert H, Jackson B, Tang SS, Schoen FJ, Smits JF, Apstein CS, Lorell BH. Distribution and functional significance of cardiac angiotensin converting enzyme in hypertrophied rat hearts. Circulation. 1993 Apr;87(4):1328-39. doi: 10.1161/01.cir.87.4.1328. PMID 8384939
- [Background] Fielitz J, Hein S, Mitrovic V, Pregla R, Zurbrugg HR, Warnecke C, Schaper J, Fleck E, Regitz-Zagrosek V. Activation of the cardiac renin-angiotensin system and increased myocardial collagen expression in human aortic valve disease. J Am Coll Cardiol. 2001 Apr;37(5):1443-9. doi: 10.1016/s0735-1097(01)01170-6. PMID 11300459
- [Background] Fujisaka T, Hoshiga M, Hotchi J, Takeda Y, Jin D, Takai S, Hanafusa T, Ishizaka N. Angiotensin II promotes aortic valve thickening independent of elevated blood pressure in apolipoprotein-E deficient mice. Atherosclerosis. 2013 Jan;226(1):82-7. doi: 10.1016/j.atherosclerosis.2012.10.055. Epub 2012 Nov 2. PMID 23177972
- [Background] Litwin SE, Katz SE, Weinberg EO, Lorell BH, Aurigemma GP, Douglas PS. Serial echocardiographic-Doppler assessment of left ventricular geometry and function in rats with pressure-overload hypertrophy. Chronic angiotensin-converting enzyme inhibition attenuates the transition to heart failure. Circulation. 1995 May 15;91(10):2642-54. doi: 10.1161/01.cir.91.10.2642. PMID 7743628
- [Background] Dahlof B, Pennert K, Hansson L. Reversal of left ventricular hypertrophy in hypertensive patients. A metaanalysis of 109 treatment studies. Am J Hypertens. 1992 Feb;5(2):95-110. doi: 10.1093/ajh/5.2.95. PMID 1532319
- [Background] Diez J, Querejeta R, Lopez B, Gonzalez A, Larman M, Martinez Ubago JL. Losartan-dependent regression of myocardial fibrosis is associated with reduction of left ventricular chamber stiffness in hypertensive patients. Circulation. 2002 May 28;105(21):2512-7. doi: 10.1161/01.cir.0000017264.66561.3d. PMID 12034658
- [Background] CONSENSUS Trial Study Group. Effects of enalapril on mortality in severe congestive heart failure. Results of the Cooperative North Scandinavian Enalapril Survival Study (CONSENSUS). N Engl J Med. 1987 Jun 4;316(23):1429-35. doi: 10.1056/NEJM198706043162301. PMID 2883575
- [Background] Greenberg B, Quinones MA, Koilpillai C, Limacher M, Shindler D, Benedict C, Shelton B. Effects of long-term enalapril therapy on cardiac structure and function in patients with left ventricular dysfunction. Results of the SOLVD echocardiography substudy. Circulation. 1995 May 15;91(10):2573-81. doi: 10.1161/01.cir.91.10.2573. PMID 7743619
- [Background] Dalsgaard M, Iversen K, Kjaergaard J, Grande P, Goetze JP, Clemmensen P, Hassager C. Short-term hemodynamic effect of angiotensin-converting enzyme inhibition in patients with severe aortic stenosis: a placebo-controlled, randomized study. Am Heart J. 2014 Feb;167(2):226-34. doi: 10.1016/j.ahj.2013.11.002. Epub 2013 Nov 9. PMID 24439984
- [Background] Bull S, Loudon M, Francis JM, Joseph J, Gerry S, Karamitsos TD, Prendergast BD, Banning AP, Neubauer S, Myerson SG. A prospective, double-blind, randomized controlled trial of the angiotensin-converting enzyme inhibitor Ramipril In Aortic Stenosis (RIAS trial). Eur Heart J Cardiovasc Imaging. 2015 Aug;16(8):834-41. doi: 10.1093/ehjci/jev043. Epub 2015 Mar 21. PMID 25796267
- [Background] Bang CN, Greve AM, Kober L, Rossebo AB, Ray S, Boman K, Nienaber CA, Devereux RB, Wachtell K. Renin-angiotensin system inhibition is not associated with increased sudden cardiac death, cardiovascular mortality or all-cause mortality in patients with aortic stenosis. Int J Cardiol. 2014 Aug 20;175(3):492-8. doi: 10.1016/j.ijcard.2014.06.013. Epub 2014 Jun 28. PMID 25012498
- [Background] Nadir MA, Wei L, Elder DH, Libianto R, Lim TK, Pauriah M, Pringle SD, Doney AD, Choy AM, Struthers AD, Lang CC. Impact of renin-angiotensin system blockade therapy on outcome in aortic stenosis. J Am Coll Cardiol. 2011 Aug 2;58(6):570-6. doi: 10.1016/j.jacc.2011.01.063. PMID 21798417
- [Background] Lund O, Erlandsen M, Dorup I, Emmertsen K, Flo C, Jensen FT. Predictable changes in left ventricular mass and function during ten years after valve replacement for aortic stenosis. J Heart Valve Dis. 2004 May;13(3):357-68. PMID 15222281
- [Background] Gjertsson P, Caidahl K, Farasati M, Oden A, Bech-Hanssen O. Preoperative moderate to severe diastolic dysfunction: a novel Doppler echocardiographic long-term prognostic factor in patients with severe aortic stenosis. J Thorac Cardiovasc Surg. 2005 Apr;129(4):890-6. doi: 10.1016/j.jtcvs.2004.09.004. PMID 15821660
- [Background] Yiu KH, Ng WS, Chan D, Sit KY, Wong A, Lee CW, Chum HL, Cheng WY, Pun CT, Ho KL, Chen Y, Ho LM, Kumana CR, Cheung HL, Chung MC, Lau CP, Au WK, Tse HF. Improved prognosis following renin-angiotensin-aldosterone system blockade in patients undergoing concomitant aortic and mitral valve replacement. Int J Cardiol. 2014 Dec 15;177(2):680-2. doi: 10.1016/j.ijcard.2014.09.163. Epub 2014 Oct 5. No abstract available. PMID 25449483
- [Background] Goel SS, Aksoy O, Gupta S, Houghtaling PL, Tuzcu EM, Marwick T, Mihaljevic T, Svensson L, Blackstone EH, Griffin BP, Stewart WJ, Barzilai B, Menon V, Kapadia SR. Renin-angiotensin system blockade therapy after surgical aortic valve replacement for severe aortic stenosis: a cohort study. Ann Intern Med. 2014 Nov 18;161(10):699-710. doi: 10.7326/M13-1505. PMID 25402513
- [Background] Dahl JS, Videbaek L, Poulsen MK, Pellikka PA, Veien K, Andersen LI, Haghfelt T, Moller JE. Effect of candesartan treatment on left ventricular remodeling after aortic valve replacement for aortic stenosis. Am J Cardiol. 2010 Sep 1;106(5):713-9. doi: 10.1016/j.amjcard.2010.04.028. Epub 2010 Jul 23. PMID 20723651
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Derived] Amat-Santos IJ, Lopez-Otero D, Nombela-Franco L, Peral-Disdier V, Gutierrez-Ibanes E, Jimenez-Diaz V, Munoz-Garcia A, Del Valle R, Regueiro A, Ibanez B, Romaguera R, Cuellas Ramon C, Garcia B, Sanchez PL, Gomez-Herrero J, Gonzalez-Juanatey JR, Tirado-Conte G, Fernandez-Aviles F, Raposeiras-Roubin S, Revilla-Orodea A, Lopez-Diaz J, Gomez I, Carrasco-Moraleja M, San Roman JA. Ramipril After Transcatheter Aortic Valve Implantation in Patients Without Reduced Ejection Fraction: The RASTAVI Randomized Clinical Trial. J Am Heart Assoc. 2024 Oct;13(19):e035460. doi: 10.1161/JAHA.124.035460. Epub 2024 Sep 18. PMID 39291483
- [Derived] Amat-Santos IJ, Santos-Martinez S, Lopez-Otero D, Nombela-Franco L, Gutierrez-Ibanes E, Del Valle R, Munoz-Garcia E, Jimenez-Diaz VA, Regueiro A, Gonzalez-Ferreiro R, Benito T, Sanmartin-Pena XC, Catala P, Rodriguez-Gabella T, Delgado-Arana JR, Carrasco-Moraleja M, Ibanez B, San Roman JA. Ramipril in High-Risk Patients With COVID-19. J Am Coll Cardiol. 2020 Jul 21;76(3):268-276. doi: 10.1016/j.jacc.2020.05.040. Epub 2020 May 26. PMID 32470515
- [Derived] Rodriguez-Gabella T, Catala P, Munoz-Garcia AJ, Nombela-Franco L, Del Valle R, Gutierrez E, Regueiro A, Jimenez-Diaz VA, Ribeiro HB, Rivero F, Fernandez-Diaz JA, Pibarot P, Alonso-Briales JH, Tirado-Conte G, Moris C, Diez Del Hoyo F, Jimenez-Britez G, Zaderenko N, Alfonso F, Gomez I, Carrasco-Moraleja M, Rodes-Cabau J, San Roman Calvar JA, Amat-Santos IJ. Renin-Angiotensin System Inhibition Following Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2019 Aug 6;74(5):631-641. doi: 10.1016/j.jacc.2019.05.055. PMID 31370954
- [Derived] Amat-Santos IJ, Catala P, Diez Del Hoyo F, Fernandez-Diaz JA, Alonso-Briales JH, Del Trigo M, Regueiro A, Juan-Salvadores P, Serra V, Gutierrez-Ibanes E, Munoz-Garcia AJ, Nombela-Franco L, Sabate M, Jimenez-Diaz VA, Garcia Del Blanco B, Lopez J, Varela-Falcon LH, Sevilla T, Arnold R, Revilla A, San Roman JA. Impact of renin-angiotensin system inhibitors on clinical outcomes and ventricular remodelling after transcatheter aortic valve implantation: rationale and design of the RASTAVI randomised multicentre study. BMJ Open. 2018 Feb 13;8(2):e020255. doi: 10.1136/bmjopen-2017-020255. PMID 29440218